CLINICAL TRIAL: NCT06602115
Title: Noncontrast CT-Based Deep Learning for Predicting Hematoma Expansion Risk in Patients with Spontaneous Intracerebral Hemorrhage
Acronym: NCCT-DL-HE
Status: Not yet recruiting | Type: Observational
Sponsor: Qiang Yu (Other)
Collaborators: Xiangya Hospital of Central South University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Southwest Hospital, China (Other); Liuzhou Workers' Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Qiang Yu, Sponsor-Investigator, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: K2023-138; K2023-138 (Other: Medical Research Ethics Committee of the First Affiliated Hospital of Chongqing Medical University)
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Spontaneous Intracerebral Hemorrhage; Hematoma Expansion
Keywords: Spontaneous Intracerebral Hemorrhage; Hematoma Expansion; Deep Learning
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (2):
- Hematoma Expansion Group: Hematoma Expansion Group
  Interventions: Other: Observational study, no interventions involved
- No Hematoma Expansion Group: Patients without hematoma expansion as defined in the study
  Interventions: Other: Observational study, no interventions involved

INTERVENTIONS:
Other: Observational study, no interventions involved — Observational study, no interventions involved

SUMMARY:
Hematoma expansion is an independent predictor of poor prognosis and early neurological deterioration in patients with spontaneous intracerebral hemorrhage. Early identification of high-risk patients and timely targeted medical interventions may provide a crucial opportunity to limit hematoma growth and improve neurological outcomes. This study aims to develop an end-to-end deep learning model based on noncontrast computed tomography images to predict the risk of hematoma expansion in patients with spontaneous intracerebral hemorrhage. This model could serve as a valuable risk stratification tool for patients with hematoma expansion, facilitating targeted treatment and providing clinicians with streamlined decision-making support in emergency situations.

DETAILED DESCRIPTION:
This project is planned to be implemented in four steps:

1. Data Collection

1. Selection of Study Subjects: Clinical and imaging data of patients with spontaneous intracerebral hemorrhage were retrospectively collected from multiple centers, including 500 cases in the hematoma expansion group and 1500 cases in the non-expansion group, totaling 2000 cases. Hematoma expansion (rHE) was defined as an absolute increase in ICH volume of ≥6 mL or a relative increase of ≥33%.
2. Collection of Clinical Data: Includes patient age, gender, history of coronary heart disease, smoking, alcohol, hypertension, admission systolic and diastolic blood pressures, among others.
3. CT Image Acquisition: Admission and follow-up CT images were obtained using spiral CT scanning with a slice thickness and interslice spacing of 5 mm.

2. Segmentation of Hematoma Based on Non-contrast CT Images Two radiologists independently segmented the volume of interest of the entire brain hematoma lesion using ITK-SNAP software, manually outlining the lesion on each CT slice while avoiding the surrounding edema and normal brain tissue.

3. Establishment of Automatic Hematoma Segmentation Model

1. Data Acquisition and Preprocessing: All images were obtained through the PACS system and stored in DICOM format. Standardized preprocessing steps were applied, including image resampling, window width, and window level adjustments to accommodate parameter differences across different CT scanners.
2. Selection of Automatic Segmentation Model: Suitable deep learning architectures for segmentation were explored and selected, including encoder-decoder structures such as nnU-Net, UNETR, and nnFormer. The optimal image segmentation model was chosen to achieve precise segmentation of brain hematoma regions.
3. Model Training and Evaluation: The model was trained using supervised learning, with manually segmented masks from the annotated dataset serving as ground truth labels. Model performance was evaluated on validation and independent external test sets using metrics such as Dice coefficient, Intersection over Union (IoU), precision, and recall.

4. Establishment of Automatic Classification Model for Hematoma Expansion

1. Construction of the Automatic Classification Model: Based on the segmentation masks extracted by the automatic segmentation model, a deep learning classification model was developed to predict hematoma expansion. Various 2D and 3D classification neural networks, including 2D-ResNet-101, 2D-ViT, 3D-ResNet-101, and 3D-ViT, were developed. Using the 3D masks generated by automatic segmentation, the largest 2D rectangular region of interest and the smallest 3D bounding box of the brain hematoma were cropped from the original CT images, and these cropped regions were input into the corresponding deep learning classification models to achieve precise prediction of hematoma expansion.
2. Visualization of the Automatic Classification Model: To visually verify the decision-making process of the deep learning model, Gradient-weighted Class Activation Mapping (Grad-CAM) technology was used to generate 2D attention maps, visually displaying the key hematoma regions identified by the model for classification.
3. Model Training and Evaluation: During model evaluation, the performance of the model was tested using an independent external test set, with comprehensive evaluation metrics including accuracy, sensitivity, specificity, F1 score, ROC curve, and AUC value. This process aimed to validate the model's generalizability and robustness across multicenter data, ensuring its reliability and effectiveness in actual clinical applications.

ELIGIBILITY:
Inclusion Criteria:

1. Primary, spontaneous (non-traumatic) intracerebral hemorrhage (ICH).
2. Age ≥ 18 years.
3. Baseline CT performed within 24 hours of ICH symptom onset or last seen well (LSW).
4. Follow-up CT within 72 hours.

Exclusion Criteria:

1. Secondary ICH caused by trauma, vascular anomalies (e.g., aneurysm, cavernous angioma, arteriovenous malformation), brain tumor, or hemorrhagic transformation in brain infarction.
2. Primary intraventricular hemorrhage (IVH).
3. Surgical treatment with external ventricular drain placement or craniotomy.
4. Obvious artifacts observed in CT images.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A multicenter retrospective cohort of 2000 patients with spontaneous intracerebral hemorrhage, including 500 cases of hematoma expansion and 1500 cases without hematoma expansion.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-09-25 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Prediction of Hematoma Expansion | From the onset of ICH symptoms to 72 hours after baseline CT
  Proportion of patients with hematoma expansion

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tran AT, Zeevi T, Haider SP, Abou Karam G, Berson ER, Tharmaseelan H, Qureshi AI, Sanelli PC, Werring DJ, Malhotra A, Petersen NH, de Havenon A, Falcone GJ, Sheth KN, Payabvash S. Uncertainty-aware deep-learning model for prediction of supratentorial hematoma expansion from admission non-contrast head computed tomography scan. NPJ Digit Med. 2024 Feb 6;7(1):26. doi: 10.1038/s41746-024-01007-w. PMID 38321131